CLINICAL TRIAL: NCT02685202
Title: The Course of Temporomandibular Pain in Response to Mandibular Advancement Therapy Among Adults With Temporomandibular Disorder and Obstructive Sleep Apnea
Brief Title: Temporomandibular Disorder (TMD) Pain in Response to Jaw Advancement in People With TMD and Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding depleted
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-4598
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Myalgia; Apnea, Obstructive Sleep
Keywords: orofacial pain; sleep-disordered breathing; temporomandibular disorder; oral appliance; upper airway collapse
MeSH Terms: conditions — Myalgia; Sleep Apnea, Obstructive; Facial Pain; Sleep Apnea Syndromes; Temporomandibular Joint Disorders | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mandibular advancement splint (Experimental): An oral appliance which is standard of care in treating mild or moderate obstructive sleep apnea by repositioning the mandible in a forward position
  Interventions: Device: Mandibular advancement splint

INTERVENTIONS:
Device: Mandibular advancement splint — A mandibular advancement splint (MAS), functions by comfortably positioning the patient's mandibular in a forward position, clearing the obstructed airway during sleep.

SUMMARY:
The purpose of this study is to characterize the course of temporomandibular disorder (TMD) pain in adults with TMD and obstructive sleep apnea (OSA), all of whom are being treated with mandibular advancement splint (MAS) therapy.

Study participants are 12 adults with painful TMD and comorbid mild to moderate OSA (apnea-hypopnea index ≥5 and <30).

This is an interventional study in which 12 patients receive MAS therapy for comorbid TMD/OSA for 16 weeks. It is standard of care to treat mild or moderate OSA with MAS therapy, the the effect on MAS therapy on TMD pain in people with OSA is unknown. There is no comparison group. Care is being provided under the direction of a sleep physician by a dentist who specializes in dental sleep medicine. The investigators expect that as MAS therapy reduces the severity of OSA, painful TMD symptoms will also reduce.

DETAILED DESCRIPTION:
Two chronic health conditions are treated with oral appliances during sleep. One condition is temporomandibular disorder (TMD); a musculoskeletal disorder characterized by pain in the masseter muscle and temporomandibular joint. TMD pain is treated with a stabilization splint which operates by limiting abnormal muscle activity. The other condition is obstructive sleep apnea (OSA). Mild to moderate OSA is treated with a mandibular advancement splint (MAS) which holds the mandible in a protruded position to increase the pharyngeal airway space and reduce upper airway collapsibility.

The comorbidity of the two conditions is high. Approximately one in four patients with clinically diagnosed TMD has OSA diagnosed by polysomnogram (PSG). This comorbidity poses a problem for management because neither appliance is considered effective in treating both conditions. In fact, mandible advancement is assumed to worsen TMD pain. However this assumption is not well supported by scientific evidence, with some studies finding that mandibular advancement actually reduces TMD pain, albeit after a transient increase in TMD pain in some patients. Furthermore, anecdotal evidence suggests that mandibular advancement reduces TMD pain. It is believed that by maintaining an open airway with the oral appliance, patients no longer have to clench their teeth in an effort to prevent the airway from collapsing during sleep.

The overall objective of this study is to characterize the temporal nature of TMD pain in adults with comorbid TMD/OSA treated with MAS therapy. It is the first study to monitor adherence to MAS therapy objectively in this study population, using a microsensor embedded in the MAS.

Recruitment and MAS therapy will be conducted at Lane and Associates Family Dentistry; a group of 27 dental practices located throughout the Triangle and Triad region of North Carolina. Advantages of using Lane & Associates are: large influx of new dental patients every month, fast recruitment, well-established protocols for screening for TMD and OSA and for referral of patients to sleep physicians for evaluation and PSG, standardized protocols for oral appliance therapy, and a Dental Sleep Medicine director who is highly experienced also in the management of TMD. The study coordinator is a dental hygienist in the University of North Carolina (UNC) School of Dentistry Dental Sleep Clinic who works in the School's Dental Sleep Medicine practice. She will travel to the Lane & Associates offices to assist in clinical and administrative activities and will manage all data collection for the 12 subjects. The Dental Sleep Clinic at the UNC School of Dentistry is not considered adequate to serve as the study site because it currently operates only one day a week and accepts referrals for only patients without TMD pain.

In the pre-enrollment phase, patients at Lane and Associates Family Dentistry will complete a standard TMD screening questionnaire. Those screening positive will be clinically examined against Research Diagnostic Criteria for TMD to confirm Group II: Masticatory Muscle Disorders, 1A: Myalgia. They will also be screened for OSA using the validated STOP-BANG questionnaire. Those at high risk will be referred for evaluation by a sleep physician and a diagnostic PSG, as is the standard of care at Lane and Associates. If the PSG reveals mild to moderate OSA (apnea-hypopnea index (AHI) ≥5 and <30), the patient is a candidate for oral appliance therapy, pending confirmation of the sleep physician, and thus eligible to enroll in the study.

Subjects will be consented and assessed for demographics, medical history, and medication use. Impressions of the upper and lower dental arches will be recorded, poured in dental stone and sent to the lab. A George Gauge will record a protrusive bite registration with the jaw advanced 60% from the most retruded position. The custom-made MAS will be fitted with a micro-recorder (Braebon DentiTrac Monitor) to assess adherence. The investigators define adherence as use of the splint 4 hours/night for ≥70% of nights as is standard practice for continuous positive airway pressure (CPAP) therapy. Home sleep test (HST): Subjects will complete a series (from 2 to 5) two-night home sleep tests (HSTs) using the portable AccuSom device by NovaSom, which collects sleep parameters of AHI, minimum oxygen saturation, and snoring indices. Novosom arranges shipment of the device and offers 24-hour technical support during the sleep test. Sleep data are uploaded wirelessly from the recorder to an online portal for statistical analysis.

Following a baseline home sleep test (HST), 12 participants will enter the study wearing a MAS during sleep that protrudes the mandible to 60% of its maximal advancement. This approximates the minimum amount of jaw advancement that is expected to be efficacious. A HST will be repeated at the end of Week #4. If that HST shows that the MAS is not efficacious (i.e. has not reduced baseline apnea hypopnea index (AHI) by ≥50% or the AHI is ≥10**), and if TMD pain is not worse, the mandible will be advanced to 70% and the participant will repeat the HST at the end of Week #8. Once efficacy is achieved, there is no need for further HSTs. If efficacy is not achieved at the end of Week #8 and if TMD pain is not worse, the mandible will be advanced to 75% and the participant will repeat the HST at the end of Week #12. If efficacy is not yet achieved and if TMD pain is not worse, the mandibular will be further advanced to 80% and the participant will undergo a final HST at the end of Week #16. Once a HST indicates that the MAS is efficacious in reducing the AHI, the participant will maintain that level of advancement. The minimum number of HSTs for any one participant is 2 (baseline and 4-week follow-up) and the maximum number is 5.

ELIGIBILITY:
Inclusion Criteria:

* Any race or ethnicity
* Meet Research Diagnostic Criteria for TMD to confirm Group II: Masticatory Muscle Disorders, 1A: Myalgia
* Rate their TMD pain severity as ≥4 on a 0-10 numeric rating scale
* Have no history of treatment for OSA.

If taking a prescription medication (with the exception of prescription formulations of NSAIDs, acetaminophen, and aspirin) episodically for the management of pain, the subject must agree to discontinue its use prior to or at the baseline visit. If taking a prescription medication daily for the management of pain, must agree to continue the daily use of the medication throughout the 16-week observation period. If taking an over-the-counter pain medication daily, the subject must agree to continue the daily use throughout the study.

Exclusion Criteria:

* <8 retained teeth per arch
* Tooth mobility
* Unmanaged periodontal disease
* Skeletal Class III occlusion
* Central sleep apnea
* Hypoventilation syndromes
* Congestive heart failure
* Chronic obstructive pulmonary disease.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Sanders, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mandibular Advancement Splint
Started | 9
Completed | 0
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Mandibular Advancement Splint
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53. (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in the Weekly Mean Pain Index Score
Description: Weekly mean pain index is computed as the arithmetic mean of daily pain index values recorded at enrollment and then at the end of each week throughout the 16 week observation period.
  Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") multiplied by pain duration (0-100 percentage scale) where percentage refers to the percent of waking day that the participant had facial pain) as reported in the Daily Symptom Diary.
  It is computed from the weekly mean pain index (numeric rating scale 0-10), and representing the arithmetic mean of daily pain index values in the preceding 7-day period. The pain index for any given day is the product of the pain intensity score multiplied by the pain duration score, each as reported in the Daily Symptom Diary kept by the subject.
Time Frame: Baseline, 16 weeks
Population: No participants could be reached to obtain pain symptom diary information; therefore, data for this outcome measure are unavailable.
Arm/Group | Mandibular Advancement Splint
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in the Apnea Hypopnea Index (AHI)
Description: The AHI is the sum of the number of apneas and hypopneas recorded during the home sleep test per hour of recorded sleep. The AHI is used to indicate the severity of obstructive sleep apnea.
Time Frame: Baseline, 16 weeks
Population: No participants could be reached to obtain apnea and hypopneas sums; therefore, data for this outcome measure are unavailable.
Arm/Group | Mandibular Advancement Splint
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in the Epworth Sleepiness Scale (ESS) Score
Description: Daytime sleepiness will be assessed using the ESS which is based on responses to self-administered questions that assess the propensity of the subject to fall asleep in 8 everyday situations (e.g., sitting and reading, talking to someone, being stopped in traffic). Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness.
Time Frame: Baseline, 16 weeks
Population: No participants could be reached to obtain ESS scores; therefore, data for this outcome measure are unavailable.
Arm/Group | Mandibular Advancement Splint
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Following splint delivery until the end of the study (approximately 12 months).
Arm/Group | Mandibular Advancement Splint
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
All nine subjects were lost to follow-up during the 16-week observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT02685202/Prot_SAP_000.pdf